CLINICAL TRIAL: NCT00005987
Title: Autologous Transplantation for Multiple Myeloma: A Research Study of Multiple Myeloma Using Chemotherapy Plus Growth Factor Primed Peripheral Blood Stem Cells Followed by Autologous Transplantation and Post-Transplant Immunotherapy
Brief Title: Filgrastim Compared With Sargramostim Plus Chemotherapy, Peripheral Stem Cell Transplantation, and Interferon Alfa in Treating Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because treatment guidelines changed
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 1996LS137; UMN-MT-9216; UMN-MT-1992-16
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Carmustine; Cyclophosphamide; Dexamethasone; Etoposide; Filgrastim; Mitoxantrone; Interferon-alpha; sargramostim; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carmustine
Drug: cyclophosphamide
Drug: dexamethasone
Drug: etoposide
Drug: filgrastim
Drug: mitoxantrone hydrochloride
Drug: recombinant interferon alfa
Drug: sargramostim
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Colony-stimulating factors such as filgrastim and sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Interferon alfa may interfere with the growth of cancer cells. It is not yet known which treatment regimen is more effective for multiple myeloma.

PURPOSE: Randomized phase II trial to compare the effectiveness of filgrastim with that of sargramostim plus chemotherapy, peripheral stem cell transplantation, and interferon alfa in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease control and extended survival in patients with multiple myeloma when treated with either filgrastim (G-CSF) or sargramostim (GM-CSF) plus high-dose chemotherapy followed by autologous peripheral blood stem cell (PBSC) transplantation followed by interferon alfa.
* Determine whether these priming treatments induce sufficient mobilization of circulating PBSC to allow their collection by leukapheresis for subsequent use in autologous transplantation in these patients.
* Determine whether these treatments induce complete response in conjunction with rapid hematopoietic recovery and modest transplant-associated morbidity and mortality in this patient population.
* Determine whether interferon alfa, given as maintenance immunostimulatory therapy for patients achieving significant cytoreduction post transplantation, can prevent or delay malignant relapse in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: In the priming phase, patients receive cyclophosphamide IV over 2 hours on day 1, mitoxantrone IV over 1 hour daily on days 1-2, and dexamethasone IV every 12 hours beginning on day 1 for a total of 4 doses. Patients also receive sargramostim (GM-CSF) IV over 2 hours or subcutaneously (SC) daily beginning 48 hours after the last dose of mitoxantrone and continuing until completion of leukapheresis. Peripheral blood stem cells (PBSC) are collected daily on days 11-13 after neutrophil recovery.
* Arm II: In the priming phase, patients receive the same treatment as in arm I except these patients receive filgrastim (G-CSF) IV over 15 minutes or SC in place of GM-CSF.

In the transplant phase, patients who have not received prior radiotherapy receive cyclophosphamide IV over 2 hours daily on days -6 and -5 and total body irradiation twice daily on days -3 through -1. Autologous PBSC are reinfused on day 0. Patients also receive GM-CSF IV over 2 hours daily and G-CSF IV over 15 minutes daily beginning on day 0 and continuing until day 28 or until blood counts recover.

Patients who have received prior radiotherapy receive cyclophosphamide IV over 2 hours daily on days -6 through -3, carmustine IV over 1 hour on day -6, and etoposide IV over 4 hours every 12 hours for a total of 6 doses on days -6 through -4. Autologous PBSC are reinfused on day 0. Patients also receive GM-CSF IV over 2 hours daily and G-CSF IV over 15 minutes daily beginning on day 0 and continuing until day 28 or until blood counts recover.

All patients then receive interferon alfa SC 3 times weekly starting on day 28 and continuing until relapse or disease progression.

Patients may also undergo radiotherapy 5 days a week for 2 weeks for residual bony lesions measuring greater than 2 cm.

Patients are followed at days 28 and 100, and at 6, 9, 12, 18, 24, 30, and 36 months.

PROJECTED ACCRUAL: A total of 25-35 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma

  * Complete or partial remission after initial therapy OR
  * Complete or partial response to therapy after disease progression following initial therapy
  * No plasma cell leukemia (greater than 10% circulating plasma cells)
  * No advanced myeloma refractory and unresponsive to at least 2 salvage chemotherapy regimens

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* Age 65-70 years:

  * Karnofsky 80-100%
* Under 65 years:

  * Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 8 g/dL (untransfused)
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3 (untransfused)

Hepatic:

* Bilirubin less than 2.0 mg/dL
* ALT less than 3 times upper limit of normal

Renal:

* Age 65-70 years:

  * Creatinine clearance greater than 60 mL/min (if creatinine at least 1.5 mg/dL)
* Under 65 years:

  * Creatinine less than 2 mg/dL

Cardiovascular:

* Age 65-70 years:

  * LVEF at least 45%
* Under 65 years:

  * No active ischemia
  * LVEF greater than 45% by MUGA

Pulmonary:

* Age 65-70 years:

  * If history of smoking or respiratory symptoms, spirometry and DLCO must be greater than 50% of predicted
* Under 65 years:

  * FEV_1 and FVC greater than 60% predicted
  * DLCO greater than 50% of predicted

Other:

* No active or uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2000-08; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States